CLINICAL TRIAL: NCT02516670
Title: A Randomized Phase 2 Trial of Ascorbic Acid in Combination With Docetaxel in Men With Metastatic Prostate Cancer
Brief Title: Docetaxel With or Without Ascorbic Acid in Treating Patients With Metastatic Prostate Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: insufficient clinical response per DSMB
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: J15106; NCI-2015-01169 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); IRB00070691 (Other: JHM IRB); J15106 (Other: Johns Hopkins University/Sidney Kimmel Cancer Center); P30CA006973 (NIH)
Record Dates: First submitted 2015-08-04; First posted 2015-08-06 (Estimated); Results first posted 2022-08-08 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: Hormone-Resistant Prostate Cancer; Metastatic Prostate Carcinoma; Stage IV Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Ascorbic Acid; Docetaxel

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (docetaxel, ascorbic acid) (Experimental): Patients receive docetaxel IV on day 1 and ascorbic acid IV twice weekly. The first ascorbic acid treatment will be given on day 1 (same day as docetaxel). Treatment repeats every 21 days for 8 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Dietary Supplement: Ascorbic Acid; Drug: Docetaxel; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Other: Quality-of-Life Assessment
- Arm B (docetaxel, placebo) (Placebo Comparator): Patients receive docetaxel IV on day 1 and placebo IV twice weekly.The first placebo treatment will be given on day 1 (same day as docetaxel). Treatment repeats every 21 days for 8 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Docetaxel; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Other: Placebo; Other: Quality-of-Life Assessment

INTERVENTIONS:
Dietary Supplement: Ascorbic Acid — Given IV
  Other Names: 2-(1,2-dihydroxyethyl)-4,5-dihydroxy-furan-3-one; Asorbicap; C Vitamin; C-Long; Ce-Vi-Sol; Cecon; Cenolate; Cetane; Cevalin; L-Ascorbic Acid; VIT C; Vitamin C; Vitamin-C
  Arms: Arm A (docetaxel, ascorbic acid)
Drug: Docetaxel — Given IV
  Other Names: RP56976; Taxotere; Taxotere Injection Concentrate
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
Other: Placebo — Given IV
  Other Names: placebo therapy; PLCB; sham therapy
  Arms: Arm B (docetaxel, placebo)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment

SUMMARY:
This randomized phase II trial studies how well docetaxel works when given with or without ascorbic acid in treating patients with prostate cancer that has spread to other places in the body. Drugs used in chemotherapy, such as docetaxel, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Ascorbic acid (vitamin C) is a water-soluble vitamin that may help inhibit the growth of cancer cells. It is not yet known whether docetaxel works better when given with or without ascorbic acid in treating prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Have metastatic castration-resistant prostate cancer (prostate cancer progressing despite castrate levels of testosterone [< 50 ng/dL] using standard measures of progression defined by Prostate Cancer Working Group 2), are chemo-naïve for metastatic castration-resistant prostate cancer (mCRPC); patients must have symptomatic disease or visceral metastases or otherwise be eligible for docetaxel treatment per investigator judgment (e.g. for progression on imaging or rapidly rising PSA despite 2nd line hormonal treatment);

  * Note: Six cycles of prior docetaxel are allowed in hormone-sensitive disease, per Eastern Cooperative Oncology Group (ECOG) 3805 data and have been off of docetaxel for at least 12 months
* Have a pathological diagnosis of prostate carcinoma
* Patients may be receiving continuous hormonal ablation with surgical or medical castration with baseline testosterone < 50 ng/dL
* Patient may be receiving bone targeted agents
* Have evaluable disease by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 and/or Prostate Cancer Working Group 2 (PCWG2) criteria
* Have ECOG performance status 0-1
* Have an estimated life expectancy > 4 months
* Absolute neutrophil count >= 1500/mm^3
* Platelets >= 100,000/mm^3
* Hemoglobin >= 9 g/dL
* Total bilirubin =< 1.0 upper limit of normal (ULN)
* Aspartate aminotransferase (AST)(serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT)(serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x ULN
* Creatinine =< 1.6 mg/dl (for patients with > 1.6 mg/dl, calculated or measured creatinine clearance must be >= 55 mL/minute [Cockcroft-Gault])
* Men of reproductive potential and those who are surgically sterilized (i.e., postvasectomy) must agree to practice effective barrier contraception that has an expected failure rate of < 1% during and for 30 days after discontinuation of study treatment

  * If condoms are used as a barrier contraceptive, a spermicidal agent should be added to ensure that pregnancy does not occur
* Have the ability to understand, and have given written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care

Exclusion Criteria:

* Have had known active central nervous system (CNS) metastases and/or carcinomatous meningitis; subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for CNS involvement for at least one week prior to trial treatment; patients with primary brain tumors are not eligible; however, as patients are completing abiraterone therapy, they will be allowed to continue up to 10 mg/day of prednisone
* Have had prior chemotherapy for metastatic disease in castration-resistant prostate cancer (prior chemotherapy for hormone-sensitive disease, more than twelve months prior to registration, is acceptable)
* Have had had surgery within four weeks of dosing of investigational agent, excluding minor procedures (dental work, skin biopsy, etc.), celiac plexus block, and biliary stent placement
* Have had palliative radiation or biological cancer therapy within 2 weeks prior to the first dose of study drug
* Have received other investigational drugs within 28 days prior to enrollment
* Is expected to require any other form of systemic or localized antineoplastic therapy while on study
* Patients who require frequent (several times a day) monitoring of their blood glucose or patients who have recently been hospitalized for glucose control
* Are being treated with anticoagulation therapy (aspirin and nonsteroidal anti-inflammatory drugs [NSAIDS] are allowed)
* The subject requires concomitant treatment with the following inhibitors of cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP3A4):

  * Antibiotics: clarithromycin, erythromycin, telithromycin, troleandomycin
  * Antifungals: itraconzaole, ketoconazole, voriconazole, fluconazole, posaconazole
  * Antidepressants: nefazodone
  * Antidiuretic: conivaptan
  * Anti-retrovirals: delaviridine or protease inhibitors (ritonavir, indinavir, lopinavir/ritonavir, saquinavir, nelfinavir) or cobicistat-boosted antiretrovirals
  * Gastrointestinal (GI): cimetidine, aprepitant
  * Hepatitis C: boceprevir, telaprevir
  * Miscellaneous: Seville oranges, grapefruit, or grapefruit juice and/or pummelos, star fruit, exotic citrus fruits, or grapefruit hybrids
* Have uncontrolled intercurrent illness, including but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Has glucose-6-phosphate dehydrogenase (G6PD) deficiency
* Have end stage renal disease
* Has history of calcium oxalate stones
* Has history of iron overload
* Have a known history of human immunodeficiency virus (HIV) (HIV 1/2 antibodies)
* Have a know active uncontrolled hepatitis B, or hepatitis C infection

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-06-20 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-10-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Channing Paller, MD, Principal Investigator — Johns Hopkins University/Sidney Kimmel Cancer Center
Locations (6):
- United States (6):
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Anne Arundel Health System, Research Institute, Annapolis, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - University Hospitals of Cleveland Seidman Cancer Center, Cleveland, Ohio
  - Thomas Jefferson University, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Paller CJ, Zahurak ML, Mandl A, Metri NA, Lalji A, Heath E, Kelly WK, Hoimes C, Barata P, Taksey J, Garrison DA, Patra K, Milne GL, Anders NM, Nauroth JM, Durham JN, Marshall CH, Markowski MC, Eisenberger MA, Antonarakis ES, Carducci MA, Denmeade SR, Levine M. High-Dose Intravenous Vitamin C Combined with Docetaxel in Men with Metastatic Castration-Resistant Prostate Cancer: A Randomized Placebo-Controlled Phase II Trial. Cancer Res Commun. 2024 Aug 1;4(8):2174-2182. doi: 10.1158/2767-9764.CRC-24-0225. PMID 39076107

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 12 subjects were Screen fails
Period: Overall Study
Arm/Group | Arm A (Docetaxel, Ascorbic Acid) | Arm B (Docetaxel, Placebo)
Started | 34 | 16
Completed | 34 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Docetaxel, Ascorbic Acid) | Arm B (Docetaxel, Placebo) | Total
Number analyzed (Participants) | 34 | 16 | 50
Age, Continuous [Mean (Full Range); unit: years] | 70 [54 to 82] | 69 [42 to 80] | 70 [42 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 34 | 16 | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 31 | 16 | 47
  Unknown or Not Reported | 3 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 6 | 11
  White | 27 | 10 | 37
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 34 | 16 | 50

OUTCOME MEASURES:

1. Primary Outcome: Number of Participates With a Decline in Prostate-specific Antigen From Their Baseline Measurement
Description: prostate-specific antigen decline will be defined as ≥ 50% from baseline measurement
Time Frame: up to 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Docetaxel, Ascorbic Acid) | Arm B (Docetaxel, Placebo)
Number analyzed (Participants) | 34 | 16
Participants | 13 | 5

2. Primary Outcome: Number of Participants With Adverse Events
Description: Number of participants experiencing fatigue, nausea, bone pain, and anorexia as defined by CTCAE 4.0
Time Frame: Up to 30 days after the last dose of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Docetaxel, Ascorbic Acid) | Arm B (Docetaxel, Placebo)
Number analyzed (Participants) | 34 | 16
Participants
  fatigue | 25 | 11
  nausea | 17 | 6
  bone pain | 2 | 2
  anorexia | 12 | 2

3. Secondary Outcome: Average Number of Times Docetaxel Had Dose Reductions
Description: The number of dose reductions and total number of completed cycles will be summarized by study arm.
Time Frame: Up to 24 weeks
Measure: Mean (Full Range); unit: dose reductions
Arm/Group | Arm A (Docetaxel, Ascorbic Acid) | Arm B (Docetaxel, Placebo)
Number analyzed (Participants) | 34 | 16
dose reductions | 7 [1 to 256] | 9 [1 to 109]

4. Secondary Outcome: Number of Serious Adverse Events
Description: Number of serious adverse events of all types as defined by Common Terminology Criteria for Adverse Events 4.0.
  A serious adverse event is an undesirable sign, symptom, or medical condition that:
  * Results in death
  * Is life threatening
  * Requires inpatient hospitalization or causes prolongation of existing hospitalization for >24 hours
  * Results in persistent or significant disability/incapacity
  * Is a congenital anomaly/birth defect
  * Is an important medical event
Time Frame: Up to 30 days after last dose of study drug
Measure: Number; unit: events
Arm/Group | Arm A (Docetaxel, Ascorbic Acid) | Arm B (Docetaxel, Placebo)
Number analyzed (Participants) | 34 | 16
events
  grade 1 | 0 | 0
  grade 2 | 4 | 0
  grade 3 | 18 | 6
  grade 4 | 3 | 0
  grade 5 | 0 | 0

5. Secondary Outcome: Number of Participates Experiencing Serious Adverse Events (SAE)
Description: Number of serious adverse events defined as grade 3 or higher (fatigue, nausea, bone pain, and anorexia) in participates as defined by CTCAE 4.0
Time Frame: Up to 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Docetaxel, Ascorbic Acid) | Arm B (Docetaxel, Placebo)
Number analyzed (Participants) | 34 | 16
Participants
  fatigue | 0 | 0
  nausea | 0 | 0
  bone pain | 0 | 0
  anorexia | 1 | 0

6. Secondary Outcome: Change in Quality of Life (QoL) as Measured by the FACT-P Questionnaire
Description: The (FACT-P) is made up of 39 question, with the total score ranging between 0 and 156 with 0 being the best and 156 as the worst.
Time Frame: Up to course 6 of therapy (18 weeks)
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Arm A (Docetaxel, Ascorbic Acid) | Arm B (Docetaxel, Placebo)
Number analyzed (Participants) | 34 | 16
score on a scale | 116.4580 [110.5926 to 122.3235] | 113.9834 [105.1710 to 122.7958]

7. Secondary Outcome: Radiographic Progression Free Survival (rPFS)
Description: To determine the rPFS of participates that receive at least one dose of ascorbic acid compared to those who received placebo
Time Frame: Up to 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A (Docetaxel, Ascorbic Acid) | Arm B (Docetaxel, Placebo)
Number analyzed (Participants) | 34 | 16
months | 10.12 [5.85 to 14.69] | 9.97 [5.32 to NA] — The upper limit of the KM curve has not reached 50%, therefore there is no estimate for the upper confidence limit on the median.

8. Other Pre Specified Outcome: Effect of Ascorbic Acid on Docetaxel Exposure
Description: To determine whether ascorbic acid alters docetaxel exposure and compare between treatment arms, pharmacokinetics samples will be collected prior to, during, and after ascorbic acid and docetaxel infusions.
Time Frame: Up to 24 weeks
Reporting Status: Not Posted

9. Other Pre Specified Outcome: F2-isoprostanes, a Pharmacodynamic Measure of Oxidant Injury in Vivo
Description: Correlative analyses will assess the association between ascorbic acid and lipid peroxidation (F2-isoprostanes) in the two study arms, globally, and over time. Comparisons of ascorbic acid and F2-isoprostanes by study arm at cycle 1, cycle 2, cycle 4 and cycle 6, accounting for baseline measures obtained from the same patient, will be made by taking differences between post baseline and baseline values and comparing these differences between arms of the study with t-tests. Regression will also be used to assess the association between F2-isoprostane and ascorbic acid at cycle 4 and at cycle 6.
Time Frame: Up to course 6 (18 weeks)
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Peak and Trough Ascorbic Acid Levels
Time Frame: Up to 24 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 30 days after the last dose of study drug
Arm/Group | Arm A (Docetaxel, Ascorbic Acid) | Arm B (Docetaxel, Placebo)
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/16
Serious Adverse Events (participants affected / at risk) | 8/34 | 3/16
Other Adverse Events (participants affected / at risk) | 34/34 | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Docetaxel, Ascorbic Acid) (N=34) | Arm B (Docetaxel, Placebo) (N=16)
Neutrophil count decreased (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (3) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Fever (General disorders) | 1 (1) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Flank Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Hip pain
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Lung infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Atrial ﬁbrillation (Cardiac disorders) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Myocardialinfarction (Cardiac disorders) | 1 (1) | 0 (0)
Investigations - Other specify (Investigations) | 1 (1) | 0 (0) — Depressed level of consciousness
Investigations - Other specify (Investigations) | 1 (1) | 0 (0) — Neutropenia
Investigations - Other specify (Investigations) | 1 (1) | 0 (0) — COLITIS
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Docetaxel, Ascorbic Acid) (N=34) | Arm B (Docetaxel, Placebo) (N=16)
Fatigue (General disorders) | 23 (43) | 11 (27)
Abdominal pain (Gastrointestinal disorders) | 3 (4) | 1 (1)
Alkaline phosphatase increased (Investigations) | 4 (11) | 4 (5)
Alopecia (General disorders) | 18 (19) | 4 (4)
Anemia (Blood and lymphatic system disorders) | 17 (34) | 3 (6)
Aneroxia (General disorders) | 13 (19) | 2 (2)
Anxiety (Psychiatric disorders) | 2 (4) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 2 (5) | 0 (0)
back pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 1 (1)
Blurred vision (Eye disorders) | 3 (3) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (12) | 2 (6)
Bruising (Injury, poisoning and procedural complications) | 3 (5) | 0 (0)
Chest pain (General disorders) | 1 (1) | 1 (3)
chills (General disorders) | 7 (8) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 2 (4) | 0 (0)
Cold symptoms (General disorders) | 3 (3) | 0 (0)
Constipation (Gastrointestinal disorders) | 16 (27) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 1 (2)
Decreased Appetite (General disorders) | 3 (3) | 0 (0)
Dehydratin (General disorders) | 3 (5) | 0 (0)
Depression (Psychiatric disorders) | 4 (4) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 23 (43) | 1 (6)
Dizziness (General disorders) | 9 (13) | 1 (1)
Dry Mouth (Gastrointestinal disorders) | 4 (6) | 3 (4)
Dysgeusia (Nervous system disorders) | 5 (8) | 3 (5)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 1 (1)
Edema (Vascular disorders) | 7 (10) | 3 (4)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 3 (5) | 0 (0)
Fever (General disorders) | 3 (6) | 2 (2)
Flatulence (Gastrointestinal disorders) | 2 (2) | 1 (1)
Flushing (Vascular disorders) | 3 (4) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1)
Headache (Nervous system disorders) | 6 (9) | 2 (4)
Hot flashes (Vascular disorders) | 6 (8) | 4 (4)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (7) | 1 (8)
Hypertension (Vascular disorders) | 10 (28) | 3 (7)
Hypocalcemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
HypoKalemia (Metabolism and nutrition disorders) | 2 (8) | 2 (3)
Hyponatremia (Metabolism and nutrition disorders) | 5 (9) | 2 (11)
Insomnia (Psychiatric disorders) | 5 (8) | 2 (3)
Light Headedness (General disorders) | 3 (4) | 0 (0)
Lymphocyte Count Decreased (Investigations) | 10 (31) | 2 (6)
Malaise (General disorders) | 4 (5) | 2 (6)
Mucositis oral (Gastrointestinal disorders) | 7 (8) | 4 (4)
Nail changes (Skin and subcutaneous tissue disorders) | 4 (4) | 2 (2)
Nausea (Gastrointestinal disorders) | 18 (34) | 6 (7)
Neuropathy sensory (Nervous system disorders) | 9 (14) | 3 (7)
Neutropenia (Investigations) | 10 (28) | 2 (2)
Neutrophil count decreased (Investigations) | 4 (9) | 0 (0)
Nocturia (General disorders) | 3 (4) | 0 (0)
Pain (General disorders) | 7 (20) | 7 (20)
Paresthesia (Nervous system disorders) | 5 (5) | 2 (4)
Platelet count decreased (Investigations) | 3 (4) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 4 (9) | 1 (2)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 1 (1)
Tachycardia (Cardiac disorders) | 2 (2) | 1 (1)
Taste Changes (General disorders) | 3 (4) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 2 (2) | 2 (2)
Urinary incontinence (Renal and urinary disorders) | 2 (4) | 1 (1)
UTI Infection (Infections and infestations) | 2 (2) | 1 (1)
Vomiting (Gastrointestinal disorders) | 8 (12) | 2 (2)
Watering Eyes (Eye disorders) | 2 (2) | 1 (1)
Weight Gain (Investigations) | 1 (2) | 3 (4)
Weight Loss (Investigations) | 4 (7) | 1 (1)
White Blood Cell Count Decreased (Investigations) | 8 (19) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-19): https://cdn.clinicaltrials.gov/large-docs/70/NCT02516670/Prot_SAP_000.pdf